CLINICAL TRIAL: NCT00170742
Title: A Randomized, Open Label, Controlled Study on the Efficacy and Safety of Octreotide i.m. in Patients With Proliferative Diabetic Retinopathy (PDR) After Start of Laser Coagulation
Brief Title: Study to Assess the Efficacy and Safety of Monthly Octreotide Intramuscular Injections in Patients With Proliferative Diabetic Retinopathy After Lasercoagulation This Study is Not Being Conducted in the United States.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: trial stopped on Sept 24, 2007
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSMS 995 H DE 07
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2008-08-12 (Estimated); Status verified 2008-08

CONDITIONS: Proliferative Diabetic Retinopathy
Keywords: Open label,; phase III,; disease,; clinical trial,; octreotide,; proliferative diabetic retinopathy, lasercoagulation
MeSH Terms: conditions — Disease | interventions — Octreotide

INTERVENTIONS:
Drug: Octreotide, 30 mg i.m. LAR formulation

SUMMARY:
Phase III study comparing monthly octreotide i.m. in comparison to no additional treatment in patients with proliferative diabetic retinopathy after lasercoagulation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with type-I or type-II-diabetes mellitus.
2. Males or females aged 18 - 70 years.
3. Proliferative diabetic retinopathy (PDR) in at least one eye that has an ETDRS visual acuity score > 35 letters (20/200 or better), and that has no other condition that might interfere with assessment of retinopathy progression (see exclusion criterion #1).
4. Media clarity, pupillary dilation and patient cooperation sufficient to allow stereoscopic 30°, or equivalent, fundus photographs of adequate quality in at least one eye that meets criterion #3 above.
5. Starting of photocoagulation of at least one eye to treat PDR in between approximately 2 weeks prior to start of study.
6. HbA1c < 13.0% at study entry. In addition, patients must be capable of testing their blood glucose levels at home and adjusting their insulin dosage to maintain blood glucose control.
7. Systolic blood pressure < 180 mm Hg and diastolic blood pressure < 105 mm Hg at study entry.
8. Females of childbearing potential must:

   * Have a negative pregnancy test prior to study entry.
   * Be practicing acceptable birth control measures inclusive of intrauterine devices or mechanical methods (i.e., oral contraceptives, vaginal diaphragm, vaginal sponge or condom with spermicide).
9. Ability to read, understand and write German language
10. Patients must give written informed consent to participate in this study.

Exclusion Criteria:

1. Pretreatment as panretinal laser treatment other than photocoagulation which started approximately 2 weeks prior to start of study (see inclusion criteria # 5).
2. Patients in whom the only otherwise eligible eye has, in the opinion of the investigator or of the central fundus photograph reading center, a condition that might interfere with assessment of retinopathy progression, including optic atrophy, extensive healed chorioretinitis, retinopathy that appears to have regressed spontaneously (with or without traction retinal detachment), retinal vascular occlusion, retinal degeneration, or other abnormality.
3. Patients with a history of symptomatic gallstones who have not had a cholecystectomy (patients with asymptomatic cholelithiasis may be entered).
4. Patients with brittle diabetes, type-I diabetes who have frequent decompensations in their glycemic control, with recurrent ketoacidosis or hypoglycemia that significantly interferes with their lifestyle.
5. Patients with a history of severe hypoglycemia unawareness.
6. Patients with a significant medical condition, other than diabetes mellitus, which may interfere with the evaluation of safety or efficacy of the study compound (e.g., unstable angina pectoris, myocardial infarction within 3 months prior to study entry, severe renal failure, patients on renal dialysis, patients who have received a renal transplant).
7. Patients who have received any investigational drug within 4 weeks prior to study entry.
8. Patients who have received prior treatment with Sandostatin or any other somatostatin analogue.
9. History of non-compliance to medical regimens or who are considered potentially unreliable Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17
Dates: Start 2003-12; Primary Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
regression of neovascularization.

SECONDARY OUTCOMES:
Determine tolerability and safety

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Customer Information, Study Chair — Novartis AG
Locations (1):
- Novartis, Basel, Switzerland